CLINICAL TRIAL: NCT06972316
Title: Effect of Global Postural Re-education in Individuals With Text Neck Syndrome
Brief Title: Global Postural Re-education in Text Neck Syndrome
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba saeid Mohamed Ahmed Elfaky, assistant lecturer of physical therapy for basic science department Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005700
Record Dates: First submitted 2025-05-01; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Text Neck Posture
Keywords: Text Neck Syndrome; postural reeducation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: 1.Group A Global Postural Re-education (Experimental): Experimental group (A) INCLUDED 30 arm with text neck syndrome ; they will received global postural reeducation and traditional treatment, The global postural reeducation was applied 3 time /week for 4 weeks.
  Interventions: Other: The Global postural reeducation
- Experimental Group B traditional tretment (Experimental): Control group (B) INCLUDED 30 arms with text neck syndrome; they will received traditional treatment, traditional treatment was applied 3 time /week for 4 weeks.
  Interventions: Other: Traditional treatments

INTERVENTIONS:
Other: The Global postural reeducation — The Global postural reeducation (GPR) is a series of postures and gentle active movements are performed aimed at stretching shortened muscles, decompressing and aligning joints, with breath¬ing contro
  Arms: Experimental: 1.Group A Global Postural Re-education
Other: Traditional treatments — Thermotherapy (hot packs) , Dynamic neck exercises, stretching exercise and posture advice
  Arms: Experimental Group B traditional tretment

SUMMARY:
The purpose of the study is to:

Investigate if there is effect of global postural re-education in individuals with text neck syndrome.

The Global postural reeducation (GPR) is a series of postures and gentle active movements are performed aimed at stretching shortened muscles, decompressing and aligning joints, with breath¬ing control, contractions of antagonist muscles and sen¬sory integration exercises to work on proprioceptive af¬ferents and re-educate postural control The study will test the following null hypothesis There is no effect of Global postural in individuals with text neck syndrome.

DETAILED DESCRIPTION:
This study will conduct in the research laboratory section, Faculty of Physical Therapy, Cairo University. The purpose of the current study will be to investigate the effect of global postural reeducation on neck pain intensity, neck disability craniovertebral angle, shoulder angle, cervical range of motion, and cervical proprioception in individuals with text neck syndrome.

This study is a Pre- test post- test single blind randomized controlled trial.

• Subjects' selection:

A. Participants:

1. 60 Participants from both genders diagnosed by physician as TNS
2. Their age will be ranging from 18-44 years old
3. Their body mass index will be ranging from (18-25) Kg/m2
4. Their using mobile phones for more than 3-4 hours per day will assess by using The Arabic version of the smartphone addiction scale
5. Informed consent (Appendix I) will be attained from each participant after clarifying the scope and purpose of the research and ensuring them of their right to decline at any time and of the privacy of any information obtained.

B- Sample size:

The sample size was calculated using the G*Power software (version 3.0.10). F-test MANOVA within and between interaction effects was selected. Considering a power of 0.80, an α level of 0.05 (2 tailed) and effect size of 0.37; two groups and number of measurements two, a generated sample size of at least 60 subjects,30 subjects per group was required.

C. Randomization:

Concealed allocation will perform by an independent person who not involved in either recruitment or treatment of the patients. He will be use individually, sequentially numbered index cards containing the randomly assigned intervention groups (A and B) that will folded and placed in sealed, opaque envelopes. the researcher will open the envelope before the 1st session and proceeds with the treatment on the initial examination day according to the group assignment.

D. Groups:

Participants will be assigned at random into 2 equal groups. Experimental group (A) received global postural reeducation and traditional treatment.

Control group (B) received traditional treatment only, which consist of [Thermotherapy (hot packs) , Dynamic neck exercises, stretching exercise and posture advice E. Incluction critrria

1. participants with age range from 18-44 years old .
2. participants with Body mass index between (18-25) Kg/m2
3. participants using mobile phones for more than 3-4 hours per day will assess by using The Arabic version of the smartphone addiction scale (short version). F. Exclusion criteria

The subject will be excluded if they had the following:

1. Individuals with a recent history of neck or back surgery.
2. Individuals with recent history of trauma or fracture.
3. Individuals with congenital disorders of the cervical spine.
4. Individuals with any psychiatric diseases.

ELIGIBILITY:
Inclusion Criteria:

* The subject will be included if they had the following:
* diagnosed by physician as text neck syndrome
* Using mobile phones for more than 3-4 hours per day
* pain score more than 4 on the visual analog scale.

Exclusion Criteria:

* The subject will be excluded if they had the following:
* a recent history of neck or back surgery.
* recent history of trauma or fracture.
* congenital disorders of the cervical spine.
* any psychiatric diseases.

Ages: 18 Months to 44 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-02-09 (Actual); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Craniovertebral angle and shoulder angle | 3 months
  Craniovertebral angle (CVA): Is the angle formed between a horizontal line through the spinous process of C7 and a line from the tragus of the ear (Ruivo et al., 2014). angles less than 49° were considered as FHP (Mani et al., 2017).
  Shoulder angle (SA): is the angle formed at a line between the center of the humerus and spinous process of C7 and the horizontal line through the center of the humerus. SA less than 52° were considered as RSP (Ruivo et al., 2014).

CONTACTS AND LOCATIONS:
Overall Officials: Heba Heba Saeid Mohamed Ahmed, master, Study Chair — Assist. lecture faculty of physical therapy Cairo university
Locations (1):
- Dokki, Cairo, Egypt